CLINICAL TRIAL: NCT02050529
Title: Randomized Controlled Trial of Labetalol Versus Hydralazine for Severe Hypertension in Obstetric Patients at a Tertiary Care Hospital of Karachi.
Brief Title: Randomized Controlled Trial of Labetalol Versus Hydralazine for Severe Hypertension in Obstetric Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Saima Aziz Siddiqui, Assistant Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Labetalol in Severe preg HTN
Record Dates: First submitted 2014-01-29; First posted 2014-01-30 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Hypertension, Pregnancy Induced; Hydralazine Adverse Reaction; Pre-eclampsia; Pre-eclampsia Superimposed Pre-existing Hypertension
Keywords: Hypertension, Pregnancy induced; Pre-eclampsia; Eclampsia; Labetalol; Hydralazine
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Eclampsia | interventions — Labetalol; Hydralazine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Labetalol (Experimental): This group (Group A; Labetalol) receiveD intravenous(IV) labetalol manufactured by Zafa pharmaceutical, 50mg/10 ml ampoule) bolus doses administered over 2 minutes, at 10 minutes interval. Initially dose of 20 mg wAS administered, and if required repeated in increments of 40 mg,80 mg,80 mg,80 mg every 10 minutes till SBP became <160 and DBP <110 mm Hg, upto a maximum cululative dose of 300mg(total 5 bolus doses).During this time pulse and blood pressure were checked every 10 minutes.
  Interventions: Drug: Labetalol
- Hydralazine (Active Comparator): This group (Hydralazine;Group B) received intravenous Hydralazine and served control. Bolus doses of 5 mg administered over 2 minutes, at 20 minutes interval. Pulse and blood pressure were checked every 10 minutes interval. If SBP threshold of 160 mm Hg or DBP 110 mm Hg was still reached after 20 minutes, then second bolus was repeated. Similarly if after 20 minutes SBP was still ≥160 or DBP ≥110 mm Hg, then third dose was given. If SBP or DBP thresholds were still exceeded after 20 minutes then similarly 4th and 5th dose of 5 mg were given. Failure to reduce SBP<160 or DBP<110 after consecutive maximum 5 boluses(total 25 mg) was labeled as severe persistent hypertension.
  Interventions: Drug: Hydralazine

INTERVENTIONS:
Drug: Labetalol — Group A( Labetalol) will be receive intravenous labetalol bolus doses as specified in protocol summary.
  Other Names: Trandate
  Arms: Labetalol
Drug: Hydralazine — Group B(Hydralazine) will serve as control and will receive active comparator Hydralazine intravenous bolus doses as specified in summary.
  Other Names: Apresoline
  Arms: Hydralazine

SUMMARY:
Severe Hypertension in pregnancy demands urgent treatment because of high mortality & morbidity in obstetric patients. Hydralazine, the most commonly used agent, causes sudden hypo tension and tachycardia. Labetalol because of combined α and β blocking effects lacks these side effects. Most recent Cochrane systematic review on use of anti hypertensive drugs in pregnancy related hypertension, could include only four trials of comparison of Hydralazine with Labetalol. Three out of total 4, had sample size ranging from 20-60 obstetric, with total sample size ranging from 19-30. Only 2 trials reported severe persistent hypertension.This review could not conclude about comparative effects due to insufficient data and suggested that further trials should compare Hydralazine with Nifedipine or labetalol, and to report severe persistent hypertension and adverse feto-maternal effects.

OBJECTIVES:1) To compare efficacy and severe persistent hypertension after intravenous Labetalol versus Hydralazine, within maximum 5 drug boluses, in obstetric severe hypertensive patients at Civil Hospital Karachi.

2) To compare immediate adverse maternal and fetal effects in the study group. 3) Furthermore, to assess response to treatment, in terms of patient and disease characteristics.

STUDY DESIGN: Randomized controlled trial.

SETTING & DURATION OF STUDY: Gynaecology Unit I, Civil hospital Karachi, from Oct 2012 to Sep 2014

METHODS: Total one hundred eighty-four patients with, severe hypertension (systolic blood pressure(S.B.P)≥160 and/or diastolic blood pressure(D.B.P) ≥110 mm Hg) at greater than 28 weeks of pregnancy or upto 72 hours after delivery, were enrolled and randomly allocated to drug A or B. At enrollment, 94 patients were allocated to Labetalol to 96 to Hydralazine through simple randomization. Since six cases were excluded due to insufficient information( 2 from group A and 4 from group B) so finally data of 92 patients in each group was analyzed. Primary outcome measures were lowering of S.B.P to <160 mm Hg and D.B.P <110 mm Hg (efficacy)and severe persistent hypertension. In addition maternal hypo tension, tachycardia, bradycardia, adverse effect on fetal heart, still birth and neonatal bradycardia were measured.

EXPECTED OUTCOME: Efficacy, severe persistent hypertension and side effects of Labetalol versus Hydralazine, in our population were determined.

Assessment of response to Drug A and B, will help in choosing a drug for different patient and disease characteristics.

DETAILED DESCRIPTION:
Study Hypothesis:Study hypothesis is that

1. There is no difference in efficacy and severe persistent hypertension after intravenous Labetalol versus Hydralazine.
2. There is no difference in adverse maternal and fetal effects.

Patients diagnosed to have severe hypertension(on repeat measurement of BP after 15 minutes of rest), admitted in 24 hour period of emergency, meeting inclusion criteria, were included. One hundred eighty-four patients were enrolled after informed consent and randomly allocated to each treatment arm by 1:1 randomization through simple random allocation.

All eligible pregnant or post partum women with systolic blood pressure ≥160mm of Hg or diastolic BP ≥110 mm Hg, on repeat measurement after 15 minutes of rest, admitted through emergency and outpatients department, were invited for participation in the study. They were enrolled after informed consent. Drug treatment was assigned using simple random sampling.

DATA COLLECTION INSTRUMENT Data was recorded on a case report form (CRF). DOSING SCHEDULE OF DRUGS A) LABETALOL: First dose of 20 mg slow intravenously over 2 minutes, if required followed at 10 minutes intervals by subsequent doses of 40 mg,80 mg, and again 80 mg repeated twice more (total 5 doses, ,maximum cumulative dose 300 mg) till primary end point i.e Systolic blood pressure <160 mm Hg and diastolic blood pressure 110 mm Hg was reached.

B)HYDRALAZINE: First dose of 5 mg slow intravenously over 2 minutes, if required followed at 20 minutes intervals by subsequent doses of 5 mg, repeated upto a maximum of 4 more times (total 5 doses, ,maximum cumulative dose 25 mg) till primary end point i.e Systolic blood pressure <160 mm Hg and diastolic blood pressure 110 mm Hg was reached.

Group A received intravenous(IV) Labetalol, bolus doses administered over 2 minutes, at 10 minutes interval. Initially dose of 20 mg was administered, and if required repeated in increments of 40 mg,80 mg, 80 mg, 80 mg every 10 minutes till SBP was reduced <160 and DBP <110 mm Hg, upto a maximum cumulative dose of 300 mg(total 5 bolus doses).During this time pulse and blood pressure were checked every 10 minutes. Failure to reduce SBP<160 or DBP<110 with consecutive maximum 5 boluses (300mg) was labelled severe persistent hypertension.In such case patient was switched to cross over treatment with hydralazine, according to dosing schedule for group B, and consultation with critical care team((Medical /cardiovascular /critical care specialist) was sought. Blood pressure and pulse were recorded at 10 minutes interval till blood pressure was reduced below threshold levels (S.B.P<160 and diastolic <110 mm of Hg).Once this level was achieved then monitoring was continued every 15 minutes interval for two hours, every 30 minutes interval for 1 hour and thereafter at hourly interval for next 4 hours.

Group B (control) received intravenous Hydralazine bolus doses of 5 mg administered over 2 minutes, at 20 minutes interval. Pulse and blood pressure were checked every 10 minutes interval. If S.B.P of 160 mm Hg or D.B.P 110 mm Hg after 20 minutes, then second bolus was repeated. Similarly if after 20 minutes S.B.P was still ≥160 or D.B.P ≥110 mm Hg, then third dose was given. If SBP or D.B.P thresholds were still exceeded after 20 minutes then similarly 4th and 5 th dose of 5 mg were given. Failure to reduce S.B.P<160 or D.B.P<110 after consecutive maximum 5 boluses(total 25 mg) was labeled as severe persistent hypertension.Once blood pressure was reduced below threshold level, pulse and blood pressure were monitored similar to group A (Labetalol). Failure to reduce S.B.P<160 or D.B.P<110 after consecutive maximum 5 boluses(total 25 mg) was labelled as severe persistent hypertension; which was considered as treatment failure. In such case, patient was switched to cross over treatment with Labetalol according to dosing schedule for group A, and emergency consultation with critical care team (Medical /cardiovascular /critical care specialist) was sought.Pulse and blood pressure was rechecked every 10 minutes till S.B.P was reduced <160 mm Hg and D.B.P <110 mm of Hg and thereafter as stated for group A.

Our use of alternate treatment for severe persistent hypertension in both groups is keeping in line with the most recent American College of Obstetricians and Gynaecologist's committee opinion 2015 recommendation.

Critical care team had authority to intervene at anytime if they thought it was necessary to interrupt treatment protocol due to patient condition or in case of non response to cross over drug.

Cardiotocography (CTG) was done in pregnant women on admission and it was repeated 2 hour after initiation of therapy.

Primary outcome measures will be lowering of SBP<160 mm Hg and DBP <110 mm Hg in scheduled dosages of allocated treatment(primary end point of study) and severe persistent hypertension i.e treatment failure.

Secondary outcome measures were adverse drug effects i.e maternal hypotension, tachycardia, bradycardia, palpitation, headache, nausea vomiting, dizziness, bronchospasm, oliguria, adverse effect on fetal heart, and neonatal bradycardia.

In both study arms, patient's monitoring and decisions for delivery of pregnant patients were taken according to department protocol which is consistent with standard recommendations.

OPERATIONAL DEFINITIONS

1. Gestational hypertension was diagnosed with a BP of ≥140/90 mm Hg after 20 weeks of pregnancy in previously normotensive women, proven by antenatal record.

2). Preeclampsia was defined as B.P ≥ 140/90 mm Hg along with proteinuria ≥ 1+ on dipsticks in a previously normotensive, non-proteinuric woman, proven by antenatal record.

3). Chronic Hypertension was diagnosed by history of preexisting hypertension & or by detecting persistent elevation of BP≥140/90 mm Hg. prior to 20 weeks of pregnancy.

4). Severe preeclampsia was defined as BP ≥160/110 along with proteinuria≥1+ on dipstick with or without one or more of the following features i.e headache, visual disturbance, upper right quadrant/epigastric pain, pulmonary oedema, elevated alanine aminotransferase (ALT), raised creatinine, hemolysis, thrombocytopenia, intrauterine growth restriction(I.U.G.R) in a previously normotensive non proteinuric woman, proven by antenatal record.

5) Eclampsia was diagnosed by generalized tonic clonic seizures in woman with hypertensive disorder not attributable to any other cause.

6) Efficacy was defined as lowering of systolic BP to <160mm Hg and diastolic BP<110 mm Hg.

7) Severe persistent hypertension was defined by SBP ≥160 or DBP≥ 110 mm of Hg after the administration of consecutive maximum (5)doses of allocated drug treatment.

8) Maternal hypotension was defined as systolic BP <90 mm Hg or diastolic BP<60 mm Hg.

9)Maternal tachycardia was defined as heart rate >100 b/m in the absence of fever & cardiovascular disease.

10)Normal Cardiotocograph(C.T.G) was defined as having following 4 features i) Baseline heart rate 110-160 beats/minute ii) Variability>5-25 beats/minutes iii) ateast 2 accelerations of >15 b/m lasting for≥15 seconds. iv) No decelerations.

11)Adverse effect on fetal heart rate (F.H.R) was defined as i)presence of any type of deceleration without uterine contraction ii)Reduced variability<5 b/m for >40 minutes, iii) Variable & late decelerations, in the presence of uterine contractions iii) F.H.R<110 b/m or >160 b/m detected on C.T.G 2 hour after starting treatment, with a baseline normal C.T.G on admission.

12)Placental abruption was defined as clinical features of uterine tenderness with evidence of retroplacental clot at delivery.

13) Oliguria was defined as urinary output<30 ml/hr for ≥4 hours. 14) Neonatal bradycardia will be defined as heart rate<100 b/m DATA ANALYSIS: Data was entered and analyzed through Statistical package for Social Sciences Software (S.P.S.S) version 20. Continuous variables i.e age, parity, gestation, Systolic blood pressure (S.B.P),Diastolic blood pressure (D.B.P), Mean arterial pressure (M,A.P) at randomization are presented as mean ± S.D whereas mean reduction in MAP, number of boluses of antihypertensive, time to achieve blood pressure control and mean dose to achieve desired level of control, were analyzed by student's t test or Mann Whitney U test, according to normality distribution. Qualitative variables i.e severe persistent hypertension, maternal hypotension, tachycardia, bradycardia, headache, palpitation, nausea vomiting,dizziness ,oliguria, placental abruption, adverse effects on fetal heart rate, still birth, neonatal bradycardia, cesarean section, Apgar score <7 at 1 and 5 minutes and neonatal intensive care admission were analyzed by chi square and Fischer's exact test(where applicable). For analyzing adverse effect on F.H.R, patients with admission C.T.G showing fetal bradycardia <110 b/m, tachycardia >160 b/m, variability <5 b/m for >40 minutes, variable and late decelerations, were excluded. Adverse effect on F.H.R was studied on all (169)antenatal women and neonatal outcomes (Apgar, neonatal bradycardia) was studied on patients delivering within 24 hours of enrollment.

Furthermore, regression model based on predictors of age cut offs ≥35 years, weight >70 kg and gestation >34 weeks was also done for both drugs.

ELIGIBILITY:
Inclusion Criteria:

INCLUSIONS CRITERIA Pregnant or post partum patients with systolic blood pressure ≥160mm of Hg or diastolic BP ≥110 mm Hg, on repeat measurement of blood pressure after 15 minutes of rest, meeting following inclusion criteria will be included.

1. Pregnancy greater than 28 wks(gestational age determined by ultrasound prior to 20 weeks which if unavailable then by uterine size at first prenatal visit or by last menstrual period) with gestational hypertension, severe preeclampsia, chronic hypertension, chronic hypertension with superimposed preeclampsia, eclampsia and unclassified hypertension.
2. Postpartum patients, upto 72 hours after delivery, diagnosed as gestational hypertension, severe preeclampsia, chronic hypertension, chronic hypertension with superimposed preeclampsia, eclampsia and unclassified hypertension.
3. Patients with singleton or multiple pregnancy.
4. Patients of all ages and parity.

Exclusion Criteria:

1. Patients with asthma.
2. Patients with cardiac failure and heart block.
3. Patients with pacing device in place or any type of cardiac arrhythmia. -

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 190 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Efficacy (Reduction in blood pressure below thresholds). | From 10 minutes upto maximum of 50 minutes from the start of Labetalol treatment (intervention arm A) and from 20 minutes up to maximum 100 minutes after start of Hydralazine treatment(control arm; B)
  Reduction in thresholds for severe hypertension in obstetric patients i.e systolic blood pressure <160 mm Hg systolic and <110 mm Hg diastolic blood pressure, with allocated drug treatment protocol and specified bolus dosages in the intervention and control(Active comparator) arms.

SECONDARY OUTCOMES:
Maternal tachycardia | Within 120 minutes of administration of any allocated drug bolus.
  Maternal tachycardia will be defined as maternal heart rate =>100 beats/min developing within 120 minutes of administration of any allocated drug bolus. After the beginning of therapy heart rate will be monitored every 10 minutes during administration of drug boluses and every15 minutes within first 2 hours of last intravenous bolus of drug in both arms.
Bradycardia | Upto 120 minutes of last intravenous drug bolus administration in both arms
  Maternal bradycardia defined as heart rate <60 beats/min developing within 120 minutes of administration of last assigned drug bolus. After the begining of therapy heart rate will be monitored every 10 minutes during administration of drug boluses and every15 minutes within first 2 hours of last intravenous bolus of drug in both arms.
Bronchospasm | Upto 120 minutes of administration of any intravenous drug bolus.
  Rhonchi developing on ausculation of chest when there was absence of Rhonchi before drug administration.
Maternal hypotension | Within 120 minutes of administration of allocated drug bolus in each arm.
  Systolic blood pressure <90 mm Hg and diastolic blood pressure < 60 mm Hg.
Adverse effect on fetal heart | 2 hours after starting treatment
  Any of the following features on cardiotocograph (C.T.G) trace, 2 hour after starting treatment, with a normal baseline C.T.G on admission.
  i) Presence of any type of deceleration without uterine contractions ii) Reduced variability<5 b/m for >40 minutes, iii) Persistent variable and late decelerations iii) Baseline fetal heart rate (F.H.R)<110b/m or >160b/m any of the following features on cardiotocography (CTG) tracing, 2 hour after starting treatment, with a normal CTG on admission. ,30, 31 i) Presence of any type of deceleration without uterine contractions ii) Reduced variability<5 b/m for >40 minutes, iii) Persistent variable and late decelerations iii) Baseline fetal heart rate (F.H.R)<110b/m or >160b/m was defined by any of the following features on cardiotocography (CTG) tracing, 2 hour after starting treatment, with a normal CTG on admission. ,30, 31 i) Presence of any type of deceleration without uterine contractions ii) Reduced variability<5 b/m for >40 minu

CONTACTS AND LOCATIONS:
Overall Officials: Saima A Siddiqui, MCPS,FCPS, Principal Investigator — Dow University of Health Science Karachi; Nazeer Khan, PhD, Study Director — Dow University of Health Health Sciences
Locations (1):
- Civil Hospital Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No